CLINICAL TRIAL: NCT06423664
Title: Pilot Feasibility Trial of Improving Neurodevelopmental ouTcomes After Prenatal Cannabinoid in uTero Exposure (INTACT)
Brief Title: Improving Neurodevelopmental ouTcomes After Prenatal Cannabinoid in uTero Exposure
Acronym: INTACT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IDeA States Pediatric Clinical Trials Network (Network)
Collaborators: University of New Mexico (Other); University of Vermont (Other); Avera Research Institute (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 276534; U24OD024957 (NIH)
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Developmental Delay
Keywords: Behavioral health intervention; Prenatal substance exposure; Neurodevelopmental outcomes; Pediatric intervention; Developmental disorders; Pediatric health
MeSH Terms: conditions — Learning Disabilities; Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: A single-arm pilot study to assess feasibility of study procedures.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Personalized coaching sessions (Experimental): A novel program to train birthing parents in contingent responding with the goal of improving neurodevelopmental outcomes in infants prenatally exposed to cannabinoids. 1 personalized coaching session per month for 12 months.
  Interventions: Behavioral: Play and Learn Strategies (PALS) Program

INTERVENTIONS:
Behavioral: Play and Learn Strategies (PALS) Program — Monthly modules and personalized coaching sessions designed to strengthen maternal responsiveness and sensitivity which, in turn, improves infant social-emotional behavior and development outcomes.
  Other Names: ePALS

SUMMARY:
The INTACT trial is a multisite pilot feasibility study aimed at testing the effectiveness of the INTACT Intervention program in improving neurodevelopmental outcomes in infants prenatally exposed to cannabinoids. The trial will enroll 20 birthing parent/infant dyads across three sites and will evaluate feasibility endpoints rather than clinical outcomes. The study duration is 22 months, including study start-up, enrollment and intervention, and data analysis and manuscript preparation.

DETAILED DESCRIPTION:
The INTACT trial is designed to address the need for interventions to improve neurodevelopmental outcomes in infants exposed to cannabinoids in utero. It is a multi-site pilot study conducted across three Institutional Development Award (IDeA) States Pediatric Clinical Trials Network (ISPCTN) sites. The trial aims to evaluate the feasibility of the INTACT Intervention program, which focuses on training birthing parents in contingent responding to promote early language, cognitive, and social development in their infants.

The study intervention consists of 12 monthly INTACT intervention coaching sessions, each comprising online module completion followed by personalized coaching sessions with interventionists certified to deliver the Play and Learn Strategies (PALS) methodology, which forms the basis for the INTACT intervention. The online modules focus on strengthening effective parenting practices, while the coaching sessions guide birthing parents in contingent responding techniques, such as reading infant signals and responding with warm and sensitive behaviors. There are three objectives for this study, examining 1) Participant Recruitment, 2) Participant Completion, and 3) Participant Adherence.

Objective 1 examines if birthing parents can be recruited and enrolled in the study. The endpoint of this objective is the percentage of potential participants approached for the study that are consented and determined to be eligible for study participation.

Objective 2 evaluates participant completion, as measured by the percent of birthing parent/infant dyads that complete the coaching session scheduled when the child is 12 months of age.

Objective 3 evaluates the number of individual INTACT intervention coaching sessions completed.

The study duration is planned for 22 months, including 1-4 months for study development and start-up, 3 months for enrollment, 12 months for the intervention, and 3 months for data organization, clean-up, and manuscript preparation.

The INTACT trial will not assess clinical outcomes but will inform the design of a future larger-scale clinical trial to evaluate the effectiveness of the INTACT Intervention program in improving neurodevelopmental outcomes in infants prenatally exposed to cannabinoids.

ELIGIBILITY:
Inclusion Criteria:

Birthing Parent

* Age of majority, as defined by the state of residency
* Cannabinoid use during pregnancy confirmed with self-report
* Have the ability to speak, read, and understand English
* Birthing parent who delivered at one of the hospitals where study team members have clinical privileges to access medical records
* Has parental custody of the infant
* Singleton pregnancy with live birth
* Has an electronic device capable of watching videos and able to stream/download videos for viewing and permitting video conferencing
* Has study access to the internet

Infant

* Term infants at birth (>37 weeks' gestation)
* Biological child of the birthing parent

Exclusion Criteria:

Birthing Parent

* Other illicit drug use, excluding cannabinoids, during pregnancy (such as heroin or cocaine) per self-reported or toxicology results
* Opiate use (prescribed or unprescribed) per self-report or toxicology results during this pregnancy
* Prolonged hospitalization following delivery longer than 7 days

Infant

* Has major birth defect(s) including physical anomalies including limb malformations/absence of limbs or chromosomal abnormalities
* Diagnosed with neonatal encephalopathy, metabolic disorder, stroke, intracranial hemorrhage, or meningitis during birth hospitalization
* Received any major surgical intervention during the birth hospitalization or required a prolonged birth hospitalization (prolonged hospitalization being any hospitalization longer than 7 days)

Max Age: 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of approached participants that are eligible for study participation | 3 months
  Whether a potential participant approached for study participation will eventually be consented and determined to be eligible for study participation.
Percentage of participants that complete their final visit | 12 months following enrollment
  Whether a birthing parent/infant dyad will complete the final coaching session when the child is 12 months of age.
Percentage of participants that receive a sufficient number of coaching sessions | 12 months following enrollment
  Whether a participant will complete the sufficient number of INTACT intervention coaching sessions, defined as completion of at least 8 out of 12 coaching sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Jessie Maxwell, MD, Principal Investigator — University of New Mexico; Leigh-Anne Cioffredi, MD, Principal Investigator — University of Vermont; Maria Barber, DO, Principal Investigator — Avera Research Institute
Locations (3):
- United States (3):
  - University of New Mexico Health Sciences Center, Albuquerque, New Mexico
  - Avera Research Institute, Sioux Falls, South Dakota
  - University of Vermont Medical Center, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
We will conduct this trial in accordance with the following publication and data sharing policies and regulations:
  NIH Public Access Policy. It requires scientists to submit final peer-reviewed journal manuscripts that arise from NIH funds to the digital archive PubMed Central upon acceptance for publication.
  ECHO ISPCTN Publications and Presentations Policy. It ensures accurate, responsible, and efficient communication of findings from ECHO ISPCTN clinical trials.
  NIH Data Sharing Policy and the policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Resulting Information Submission Rule. Other researchers may request data from this trial by contacting Song Ounpraseugh, PhD, at the ISPCTN Data Coordinating and Operations Center (DCOC).
Supporting Information: SAP, ICF
Time Frame: Per data sharing polices of NIH and the ISPCTN
Access Criteria: to be announced

REFERENCES:
- [Derived] Maxwell JR, Cioffredi LA, Talavera-Barber MM, Henry M, Beauman S, Hittson A, McCoy M, Chassereau L, Jin J, Abraham PA, Fu LY, Raissy H, Snowden JN. The protocol for a pilot feasibility trial of Improving Neurodevelopmental ouTcomes After prenatal Cannabinoid in uTero exposure (INTACT) study for a multi-center trial. PLoS One. 2025 May 12;20(5):e0322035. doi: 10.1371/journal.pone.0322035. eCollection 2025. PMID 40354465